CLINICAL TRIAL: NCT05554705
Title: A Lifestyle Intervention for Rheumatoid Arthritis: Effect of an Intensive Therapeutic Lifestyle Change Program on Inflammatory Markers and Clinical Outcomes
Brief Title: Lifestyle Intervention for Rheumatoid Arthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lost necessary staff support
Sponsor: Blue Cross Blue Shield of Vermont (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-08-629-1275
Record Dates: First submitted 2022-09-17; First posted 2022-09-26 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Lifestyle Risk Reduction; Rheumatoid Arthritis
MeSH Terms: conditions — Risk Reduction Behavior; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): standard of care + lifestyle intervention
  Interventions: Behavioral: Intensive Lifestyle intervention
- control (No Intervention): no intervention (control group)

INTERVENTIONS:
Behavioral: Intensive Lifestyle intervention — 12 week therapeutic lifestyle change program
  Arms: experimental

SUMMARY:
The main purpose of this study is to assess whether adding a multifaceted lifestyle intervention to the standard best practice of care can be more effective than standard best practices alone for treating Rheumatoid Arthritis.

DETAILED DESCRIPTION:
The main purpose of this study is to assess whether adding a multifaceted lifestyle intervention to the standard best practice of care can be more effective than standard best practices alone for treating Rheumatoid Arthritis. If a lifestyle intervention is effective, we expect to see improvement in functional status and decreased health care costs to the study participant and the insurer.

ELIGIBILITY:
Inclusion Criteria:

1. BCBSVT members who also carry the prescription benefit with BCBSVT (due to the need for tracking prescription costs).
2. BCBSVT membership for minimum of 12 months prior to start of study (due to the need for tracking prescription costs before and after intervention).
3. Age 18 or older
4. Medical diagnosis of RA

Exclusion Criteria:

1. Pregnancy
2. Currently taking warfarin (since fluctuating amounts of green leafy vegetable intake can adversely affect INR levels and because we will be asking participants to increase the amount of green leafy vegetables they consume)
3. Malignancy currently undergoing treatment (with further planned treatment at the time of enrollment) since patients undergoing cancer treatment often need to stop RA medications in order to improve immune function, and thus could be a confounder.
4. Food allergy (including reactions such as hives, wheezing, difficulty breathing, fainting, or anaphylaxis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Change in HAQ-2 score | Up to 24 months
  The HAQ-II is a validated and reliable tool used frequently by rheumatologists evaluating patients with RA (Wolfe et al, 2004). It is an indicator of quality of life as well as functional status. It is also a predictor of premature mortality.
Change in serum C-Reactive Protein | Up to 24 months
  CRP is a reliable marker of acute and chronic inflammation (Sproston and Ashworth, 2018).

SECONDARY OUTCOMES:
Change in dosage of RA-related medications | Up to 24 months
  Dosage of Medications Taken Specifically for Rheumatoid Arthritis
Change in the number of medications required to treat RA | Up to 24 months
  Number of Medications Taken Specifically for Rheumatoid Arthritis
Change in RA-related costs for the study participant | Up to 24 months
  Out of Pocket costs related to Rheumatoid Arthritis Care
Change in RA-related costs to the insurer | Up to 24 months
  Costs for care of Rheumatoid Arthritis paid by insurer
Change in serum LDL cholesterol | Up to 24 months
  Elevated Low Density Lipoprotein is strongly associated with heart disease
Change in serum total cholesterol | Up to 24 months
  Elevated total cholesterol is associated with heart disease
Change in serum HbA1c | Up to 24 months
  Hemoglobin HbA1c is used to assess glucose control in diabetics
Change in blood pressure | Up to 24 months
  Blood pressure change
Change in BMI | Up to 24 months
  Body Mass Index change
Change in weight | Up to 24 months
  Weight change

CONTACTS AND LOCATIONS:
Overall Officials: Keri LeCompte, PharmD, Principal Investigator — Blue Cross Blue Shield of Vermont
Locations (1):
- Blue Cross Blue Shield of Vermont, Berlin Corners, Vermont, United States

IPD SHARING:
Plan to Share IPD: No